CLINICAL TRIAL: NCT03707756
Title: Systematic Review of Phenotype Characteristics of DFNA9 Caused by the Pro51 Ser (P51S) Mutation in COCH
Brief Title: Systematic Review of Phenotypical Characteristics of P51S COCH Mutation
Status: Withdrawn | Type: Observational
Why Stopped: systematic literature review has been completed
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Sebastien Janssens de Varebeke, principal investigator, Jessa Hospital
Other Study IDs: JessaH-ORL-1
Record Dates: First submitted 2018-10-08; First posted 2018-10-16 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: DFNA9
Keywords: DFNA9; COCh; Mutation; Genotype-phenotype

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Gene mutations account for more than 60% of congenital sensorineural hearing loss (SNHL) in Western Countries. Hereditary SNHL does not necessarily start at birth, however, as many causative gene mutations only begin to express at much later ages, such as for example DFNA9, also known as the ninth discovered autosomal dominant SNHL.

It is characterized by a late onset of rapid progressive SNHL together with accompanying vestibular impairment. The first reported DFNA9 patients were carrying the c.151 C>T mutation in COCH, which is the result of a substitution of cytosine by thymine nucleotide of the 151th base pair (c.151C>T). At protein level, this missense point mutation induces a mistranslation to a serine instead of a proline amino-acid (p.Pro51Ser, (P51S)), producing mutant cochlin that cause a dominant negative effect due to misfolding.

In the perspective of promising future hearing and vestibular treatment developments, such as gene therapy, stem cell therapy, neural regeneration, in association with cochlear and/or vestibular implantation, a more accurate understanding of the onset of the very first signs of the auditory and vestibular deterioration is important. However, in early stages these first signs of impairment are very discrete and pre-symptomatic.

The aim of this systematic review is to identify studies related to DFNA9, caused by the P51S COCH variant, describing detailed genotype-phenotype correlation in relation to the age and to investigate the age of onset of the SNHL and peripheral vestibular function as well as their progression in relation to age.

DETAILED DESCRIPTION:
The strategy and methodology used for the systematic review was based on the PRISMA Statement (Preferred Reporting Items for Systematic Reviews and Meta-Analysis Medline, PubMed, Cochrane Database of Systematic Reviews, Cochrane Central Register of Controlled Trials, ISI Web of Knowledge and Web of Science were searched. Information was retrieved about COCH mutations causing DFNA9, including phenotype, genotype, audiometric and vestibular data.

Audiometric data were collected using individual measurements or pure tone average incides in the selected records.In case of different audiometric data presentation, for instance audiograms or different pure tone average (PTA) plots against age, a comprehensive assessment and inventory of all individual measurements was conducted. All available measurements at both ears per frequency were inventoried and a binaural mean value for each frequency per age was averaged, before the calculation of the indices. If longitudinal measurements of the same individual were shown, all the available data was included in the assessment.

The following parameters for the audiometric data were inventoried: pure tone average (PTA), Annual Threshold detarioration (ATD) per frequency and/or PTA, Age-related Typical Audiogram (ARTA) and age of onset of the sensorineural hearing loss (SNHL).

For the vestibular function, all different parameters of the vestibular function were inventoried. Normative values, if mentioned, were used to evaluate the measurements. An overall inventory of all individual vestibular measurements in relation to age was conducted.

The following parameters for the vestibular function were inventoried: Time Constant (T) derived from velocity-step test (VST) in seconds, Caloric response gain on electronystagmography, Annual vestibular deterioration rate and age of onset of vestibular dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* P51S carriership

Exclusion Criteria:

* no P51S carriership

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all affected subjects carrying the P51S COCH mutation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
age of onset sensorineural hearing loss | 10 years
  Age of onset sensorineural hearing loss (years) in P51S COCH mutation carriers
annual threshold deterioration | 10 years
  Annual threshold deterioration (decibel hearing loss per year) in P51S COCH mutation carriers
age of onset vestibular dysfunction | 10 years
  Age of onset vestibular dysfunction (time constant T (seconds) in P51S COCH mutation carriers
annual vestibular deterioration rate | 10 years
  Annual vestibular deterioration (seconds per year) in P51S COCH mutation carriers
Pure Tone Average (PTA) | 10 years
  Pure tone average (PTA) in decibel hearing loss (dB HL) of P51S COCH mutations carriers
Age-Related Typical Audiogram (ARTA) | 10 years
  Age-related typical audiogram (ARTA) of P51S COCH mutation carriers
Time Constant 'T' | 10 years
  Time constant 'T' with velocity-step test(VST) (seconds) in P51S COCH mutation carriers
gain of caloric test of ENG | 10 years
  summation of gain in caloric test of electronystagmography (ENG) (degrees per second) of P51S COCH mutation carriers